CLINICAL TRIAL: NCT05665504
Title: Using Biomarkers for Diagnosis, Risk Stratification of Post -Treatment Recurrence and Long-Term Surveillance of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-21767
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung; Node; Adenocarcinoma of Lung
Keywords: Biomarkers; Lung Cancer Biomarkers
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- High-Risk for Recurrence That Accept Adjuvant Chemotherapy: Participants whose gene assay show that they are at a higher risk of recurrence will be offered to receive postoperative chemotherapy. If participants also have a special mutation on the tumor (EGFR), investigators will recommend that the participant also receive the oral anti-EGFR pill (TagrissoTM) daily for 3 years after completing the chemotherapy. The administration of standard postoperative chemotherapy is not considered part of the study. Only the results of the DetermaRx test is a part of this study.
  Interventions: Diagnostic Test: DetermaRX
- High-Risk for Recurrence That Decline Adjuvant Chemotherapy: Participants whose gene assay show that they are at a higher risk of recurrence will be offered to receive postoperative chemotherapy. If participant declines, investigators will followup with participants periodically every 6-12 months over 5 years.
  Interventions: Diagnostic Test: DetermaRX
- Low-Risk for Recurrence: Participants whose gene assay show that they are at a lower risk of recurrence will not be offered additional treatment after resection. Investigators will followup with participants periodically every 6-12 months over 5 years.
  Interventions: Diagnostic Test: DetermaRX

INTERVENTIONS:
Diagnostic Test: DetermaRX — A lung tissue biomarker to risk stratify patients immediately after curative lung cancer resections into groups with low risk versus intermediate-high risk for recurrence of cancer. Intermediate-high risk patients will be advised to undergo adjuvant chemotherapy with the expectation of decreasing their chance of recurrence. The effectiveness and toxicity of the adjuvant chemotherapy itself is considered not part of the study-just the decision to recommend adjuvant chemotherapy is the study intervention. Investigators will then evaluate the long-term survival results of low-risk patients (no adjuvant treatment) and intermediate-high risk patients receiving adjuvant treatment versus intermediate-high risk patients who decline adjuvant therapy.

SUMMARY:
This study is an observational study of blood and tissue biomarkers. Investigators plan to evaluate the accuracy of lung cancer biomarkers found in the blood in determining if a lung nodule is cancer or benign. Investigators also plan to examine another biomarker found in the tumor tissue to identify participants after lung cancer surgery who have a high risk for recurrent cancer. Finally, investigators plan to determine if one of the blood-based biomarkers can be used to detect any late cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Potentially-resectable lung nodule 8-40 mm diameter suspected (no preop diagnosis) of being a clinically node-negative lung cancer [clinical stage IA-IB (cT1a-T2aN0), <4cm diameter].
* If surgical resection is recommended, patient will undergo surgery at Moffitt Cancer Center.
* If a definite tissue diagnosis is obtained and stereotactic body radiotherapy (SBRT) is the recommended treatment instead of surgery, the SBRT will be delivered at Moffitt Cancer Center.
* >18 years old, male or female.
* ECOG performance status 0-1.
* Agree to participate in the follow-up protocol.
* Any suspected primary lung cancer cell type (except a suspected typical carcinoid tumor, carcinoma in situ or minimally-invasive carcinoma).
* Ability to understand and the willingness to sign a written, informed consent document.

Exclusion Criteria:

* Participants who are actively receiving any cancer treatment.
* Participants with uncontrolled intercurrent illness.
* Prior lung cancer within 5 years.
* Current active other major cancer except non-melanoma skin cancer.
* Patients with pure ground glass opacities (nodules) or hilar masses.
* Suspected typical carcinoid cell type (well-differentiated neuroendocrine carcinoma).
* Metastatic nodule (suspected) in the lung from an extrapulmonary cancer.
* Patient unable to provide informed consent.
* Prisoner or incarcerated individual.
* For surgical patients, a R1 or R2 resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in the Moffitt Thoracic Surgery and Lung Diagnosis Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | Up to 5 years
  Disease-free survival (DFS) is defined as the time from surgical resection and adjuvant chemotherapy to recurrence of tumor or death
Overall Survival | Up to 5 Years
  Overall survival (OS) is defined as the time (days) from the date of surgical resection and adjuvant chemotherapy to the date of death, due to any reason.

SECONDARY OUTCOMES:
Tumor Malignancy | At 6 Months
  Fisher exact test will used to test association of both LCDT1™, NodifyXL2®, and CIZ1b™ blood tests with malignancy.
Cancer Recurrence | At 6 Months
  Fisher exact test will used to test association of LCDT-1™ blood test with cancer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Lary A Robinson, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Search — https://moffitt.org/clinicaltrialssearch?DiseaseSite=&q=21767&SortCriteria=